CLINICAL TRIAL: NCT00867100
Title: A Randomized, Double-blind, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 827 in Healthy Subjects and Subjects With Moderate to Severe Psoriasis
Brief Title: Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 827
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060279
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo
- 140 mg SC (Experimental): 140 mg SC PsO
  Interventions: Drug: 140 mg SC
- 350 mg SC (Active Comparator): 350 mg SC PsO
  Interventions: Drug: 350 mg SC
- 700 mg IV (Experimental): 700 mg IV PsO
  Interventions: Drug: 700 mg IV

INTERVENTIONS:
Drug: 700 mg IV — single SC or IV dose in healthy subjects (Part A) and subjects with moderate to severe psoriasis (Part B).
  Arms: 700 mg IV
Drug: 350 mg SC — single SC or IV dose in healthy subjects (Part A) and subjects with moderate to severe psoriasis (Part B).
  Arms: 350 mg SC
Drug: Placebo — single SC or IV dose in healthy subjects (Part A) and subjects with moderate to severe psoriasis (Part B).
  Arms: Placebo
Drug: 140 mg SC — single SC or IV dose in healthy subjects (Part A) and subjects with moderate to severe psoriasis (Part B).
  Arms: 140 mg SC

SUMMARY:
This Phase 1 study will evaluate safety, tolerability, PK and PD of AMG 827 when administered as a single SC or IV dose.

DETAILED DESCRIPTION:
This Phase 1 study will evaluate safety, tolerability, PK and PD of AMG 827 when administered as a single SC or IV dose in healthy subjects (Part A) and subjects with moderate to severe psoriasis (Part B).

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Able to provide written informed consent
* Healthy male or female between 18 to 45 years of age, inclusive at the time of screening
* Additional inclusion criteria apply

Part B:

* 18 - 55 years old inclusive at Screening
* Active but clinically stable, plaque psoriasis
* Psoriasis involving ≥ 10% of the body surface area
* A minimum PASI score of ≥ 10 obtained during the screening period
* Additional inclusion criteria apply

Exclusion Criteria:

Part A:

* History or evidence of a clinically significant disorder (including but not limited to cardiopulmonary, oncologic, renal, metabolic, hematologic or psychiatric), condition or disease that, in the opinion of the Investigator and Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Underlying condition that predisposes the subject to infections (eg, uncontrolled diabetes - HbA1c > 7%, history of splenectomy)
* Additional exclusion criteria apply

Part B:

* Active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit
* Evidence of skin conditions other than psoriasis (eg, eczema) at the time of the screening visit or between the screening visit and study drug initiation that would interfere with evaluations of the effect of investigational product on psoriasis
* Any condition that, in the judgment of the investigator, might cause this study to be detrimental to the subject
* Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Papp KA, Reid C, Foley P, Sinclair R, Salinger DH, Williams G, Dong H, Krueger JG, Russell CB, Martin DA. Anti-IL-17 receptor antibody AMG 827 leads to rapid clinical response in subjects with moderate to severe psoriasis: results from a phase I, randomized, placebo-controlled trial. J Invest Dermatol. 2012 Oct;132(10):2466-2469. doi: 10.1038/jid.2012.163. Epub 2012 May 24. No abstract available. PMID 22622425
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Part B; Placebo Part A: Single SC or IV dose of matching placebo
- Cohort 10: 140 mg Sc Part B: 140 mg Sc PsO Population
  Adults with Psoriasis
- Cohort 11: 350 mg Sc Part B: 350 mg Sc PsO population
  Adults with Psoriasis
- Cohort 9: 700 mg IV Part B: 700 mg IV PsO population
  Adults with Psoriasis
- Cohort 1: 7mg SC Part A: 7mg SC PsO population
- Cohort 2: 21mg SC Part A: 21mg SC PsO population
- Cohort 3: 21mg IV Part A: 21 mg IV PsO population
- Cohort 4: 70mg SC Part A: 70mg SC PsO population
- Cohort 5: 210mg SC Part A: 210mg SC PsO population
- Cohort 6: 210mg IV Part A: 210 mg IV PsO population
- Cohort 7: 420mg SC Part A: 420mg SC PsO Population
- Cohort 8: 700mg IV Part A: 700mg IV PsO population
Period: Overall Study
Arm/Group | Placebo Part B | Cohort 10: 140 mg Sc Part B | Cohort 11: 350 mg Sc Part B | Cohort 9: 700 mg IV Part B | Placebo Part A | Cohort 1: 7mg SC Part A | Cohort 2: 21mg SC Part A | Cohort 3: 21mg IV Part A | Cohort 4: 70mg SC Part A | Cohort 5: 210mg SC Part A | Cohort 6: 210mg IV Part A | Cohort 7: 420mg SC Part A | Cohort 8: 700mg IV Part A
Started | 5 | 5 | 8 | 8 | 14 | 6 | 7 | 3 | 6 | 6 | 4 | 6 | 6
Completed | 5 | 4 | 8 | 8 | 14 | 6 | 6 | 3 | 6 | 6 | 3 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 140 mg SC Part B: 140 mg Sc PsO Population
- 350 mg SC Part B: 350 mg Sc PsO population
- 700 mg IV Part B: 700 mg IV PsO population
- 7mg SC Part A: 7mg SC PsO population
- 21mg SC Part A: 21mg SC PsO population
- 21mg IV Part A: 21mg IV PsO population
- 70mg SC Part A: 70mg SC Pso population
- 210mg SC Part A: 210mg SC PsO population
- 210mg IV Part A: 210mg IV PsO population
- 420mg SC Part A: 420mg SC PsO population
- 700mg IV Part A: 700mg IV PsO population
- Total: Total of all reporting groups
Arm/Group | Placebo Part B | 140 mg SC Part B | 350 mg SC Part B | 700 mg IV Part B | Placebo Part A | 7mg SC Part A | 21mg SC Part A | 21mg IV Part A | 70mg SC Part A | 210mg SC Part A | 210mg IV Part A | 420mg SC Part A | 700mg IV Part A | Total
Number analyzed (Participants) | 5 | 4 | 8 | 8 | 14 | 6 | 6 | 3 | 6 | 6 | 4 | 6 | 6 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (6.6) | 34.5 (11.7) | 39.5 (13.4) | 43 (11.6) | 23.1 (2.5) | 25.5 (8.2) | 27.0 (8.6) | 25.3 (2.5) | 22.2 (1.5) | 28.3 (9.9) | 21.3 (2.2) | 24.5 (6.6) | 24.3 (3.0) | 32.75 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Male | 3 | 3 | 6 | 7 | 14 | 6 | 6 | 3 | 6 | 6 | 4 | 6 | 6 | 76

OUTCOME MEASURES:

1. Primary Outcome: Part B: PASI (Psoriasis Area and Severity Index) Score Mean Percentage of Change Through Day 43
Description: Summary of percent change in PASI (Psoriasis Area Severity Index) Scores over time by treatment groups between baseline and day 43, PASI score ranging from (0) no disease to (72) maximal disease.
Time Frame: Through day 43
Population: This PASI outcome measure data refers only to Part B subjects with moderate to severe plaque psoriasis.
Measure: Mean (Standard Deviation); unit: percentage improvement
Groups:
- Placebo: Placebo-treated
- 140 mg Sc: 140 mg Sc PsO Population
- 350 mg Sc: 350 mg Sc PsO population
- 700 mg IV: 700 mg IV PsO population
Arm/Group | Placebo | 140 mg Sc | 350 mg Sc | 700 mg IV
Number analyzed (Participants) | 5 | 4 | 8 | 8
percentage improvement | 19.88 (6.36) | 17.74 (15.34) | 53.57 (30.45) | 86.04 (8.70)

2. Primary Outcome: Part B: All Treatment Adverse Events Reported for Safety Evaluation
Description: This primary outcome assesses number of participants iwth any reported adverse events emerging during treatment period.
Time Frame: 85 days
Measure: Number; unit: participants with events
Groups:
- Placebo Part B: Placebo-treated
Arm/Group | Placebo Part B | 140 mg Sc Part B | 350 mg Sc Part B | 700 mg IV Part B
Number analyzed (Participants) | 5 | 4 | 8 | 8
participants with events | 4 | 3 | 7 | 8

3. Primary Outcome: Part A: All Treatment Adverse Events Reported for Safety Evaluation
Description: This primary outcome assesses the number of participants with any reported adverse events emerging during treatment period.
Time Frame: Cohort 1-4 43 days, Cohort 5-8 64 days
Measure: Number; unit: participants with events
Arm/Group | Placebo Part A | Cohort 1: 7mg SC Part A | Cohort 2: 21mg SC Part A | Cohort 3: 21mg IV Part A | Cohort 4: 70mg SC Part A | Cohort 5: 210mg SC Part A | Cohort 6: 210mg IV Part A | Cohort 7: 420mg SC Part A | Cohort 8: 700mg IV Part A
Number analyzed (Participants) | 14 | 6 | 6 | 3 | 6 | 6 | 4 | 6 | 6
participants with events | 14 | 6 | 6 | 3 | 6 | 6 | 4 | 5 | 6

ADVERSE EVENTS:
Groups:
- Cohort 10: 140 mg Sc Part B: 140 mg Sc PsO Population
- Cohort 11: 350 mg Sc Part B: 350 mg Sc PsO population
- Cohort 9: 700 mg IV Part B: 700 mg IV PsO population
- Cohort 2: 21mg SC Part A: 21mg SC PsO population ...
- Cohort 3: 21mg IV Part A: 21 mg IV PsO population ...
- Cohort 4: 70mg SC Part A: 70mg SC PsO population ...
- Cohort 5: 210mg SC Part A: 210mg SC PsO population ...
- Cohort 6: 210mg IV Part A: 210 mg IV PsO population ...
- Cohort 7: 420mg SC Part A: 420mg SC PsO Population ...
- Cohort 8: 700mg IV Part A: 700mg IV PsO population ...
Arm/Group | Placebo Part B | Cohort 10: 140 mg Sc Part B | Cohort 11: 350 mg Sc Part B | Cohort 9: 700 mg IV Part B | Placebo Part A | Cohort 1: 7mg SC Part A | Cohort 2: 21mg SC Part A | Cohort 3: 21mg IV Part A | Cohort 4: 70mg SC Part A | Cohort 5: 210mg SC Part A | Cohort 6: 210mg IV Part A | Cohort 7: 420mg SC Part A | Cohort 8: 700mg IV Part A
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/8 | 0/8 | 0/14 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 8/8 | 8/8 | 14/14 | 6/6 | 6/6 | 3/3 | 6/6 | 6/6 | 4/4 | 5/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Part B (N=5) | Cohort 10: 140 mg Sc Part B (N=4) | Cohort 11: 350 mg Sc Part B (N=8) | Cohort 9: 700 mg IV Part B (N=8) | Placebo Part A (N=14) | Cohort 1: 7mg SC Part A (N=6) | Cohort 2: 21mg SC Part A (N=6) | Cohort 3: 21mg IV Part A (N=3) | Cohort 4: 70mg SC Part A (N=6) | Cohort 5: 210mg SC Part A (N=6) | Cohort 6: 210mg IV Part A (N=4) | Cohort 7: 420mg SC Part A (N=6) | Cohort 8: 700mg IV Part A (N=6)
Conjunctival Irritation (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesphageal Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post Procedural Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Injection Site Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 6 | 5 | 6 | 0 | 1 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 7 | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrheoa (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 7 | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Koebner Phenomenon (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other